CLINICAL TRIAL: NCT06824545
Title: Incidence & Clinical Significance of Osteolysis Following PEEK Suture Anchor Use in Hand & Wrist Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 24-1667
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Osteolysis
MeSH Terms: conditions — Osteolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent hand & wrist surgery with suture anchor implantation over the past 10 years.

SUMMARY:
This prospective observational study evaluates the incidence & clinical significance of osteolysis following polyetheretherketone (PEEK) suture anchor use in hand & wrist surgery. Building on a pilot study, it focuses on patients undergoing hand & wrist surgeries with suture anchor implantation over the past 10 years. Patients are grouped by anchor composition: PEEK, metallic, or bioabsorbable. The investigators hypothesize that PEEK anchors will show significantly greater osteolysis than metallic or bioabsorbable anchors. Furthermore, among all patients with osteolysis, the investigators expect no statistically significant differences in patient-reported outcomes (PROs), post-op complications, or revision surgery rates, regardless of anchor type. Lastly, for patients with ulnar collateral ligament (UCL) thumb injuries, the investigators hypothesize that osteolysis presence will not correlate with increased UCL laxity upon valgus stress testing compared to the nonoperative thumb.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 99 years-old
* History of hand and/or wrist surgery with suture anchor fixation over the 10-year period between January 1, 2014 and January 1, 2024.
* Possess an en face and/or tangential radiograph of the suture anchor tunnels from either the intra-operative or immediately post-operative (within 14 days) period.

Exclusion Criteria:

* Systematic inflammatory / autoimmune disease or immune-modulatory drug use.
* History of revision surgery of the body part of interest.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 2014 & 2024 who were billed for one of the following CPT codes: 25310, 25320, 25447, 26480, 26540, 226541, 26542, and 26545.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Rates of Osteolysis | 18 months
  This analysis focuses on the primary outcome of osteolysis rates within the patient populations who received one of three difference suture anchor types (PEEK, bioabsorbable, or metallic) - as defined by the number of patients per anchor type presenting with >30% increases in the size of suture anchor tunnels between their immediate & final post-operative X-ray series.

CONTACTS AND LOCATIONS:
Locations (1):
- UCHealth Steadman Hawkins Clinic Inverness, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No